CLINICAL TRIAL: NCT06622421
Title: Piezoeletric Surgery vs Conventional Surgery for Treatment of Medication-related Osteonecrosis of the Jaws: a Randomized Clinical Trial
Brief Title: Piezoeletric Surgery vs Conventional Surgery for Treatment of MRONJ
Acronym: PIEZOPZ-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5786
Record Dates: First submitted 2024-07-16; First posted 2024-10-02 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-09

CONDITIONS: Bisphosphonate-Associated Osteonecrosis of the Jaw; Osteonecrosis of the Jaw; Osteonecrosis Due to Drug
Keywords: MEDICATION RELATED OSTEONECROSIS OF THE JAW; SURGICAL TREATMENT OF MRONJ; MRONJ
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized and controlled study with parallel groups (1:1) of superiority
Who Masked: Investigator, Outcomes Assessor
Masking Description: The collaborator who will collect the data and the statistician will not be aware of the assignment group. Each patient will be identified with a unique code (PIEZOPZ_n.) that will be known only to the principal investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1 - control group (Other): Patients with MRONJ diagnosis who will undergo to conventional surgery using rotary burns instruments
  Interventions: Procedure: Conventional surgery
- G2 - study group (Experimental): Patients with MRONJ diagnosed who will undergo to piezoelectric surgery
  Interventions: Device: Piezoelectric surgery

INTERVENTIONS:
Device: Piezoelectric surgery — Patients enrolled and randomized into one of the two groups will all undergo surgery to remove necrotic bone on an outpatient basis by the same operator with a decade of experience in the treatment of MRONJ. As per clinical routine, a marginal bone resection procedure will be performed using rotary instruments or piezoelectric instruments (depending on the assignment to one of the two groups). Both surgical procedures involve complete closure of the wound by primary intention using sutures
  Arms: G2 - study group
Procedure: Conventional surgery — Patients enrolled and randomized into one of the two groups will all undergo surgery to remove necrotic bone on an outpatient basis by the same operator with a decade of experience in the treatment of MRONJ. As per clinical routine, a marginal bone resection procedure will be performed using rotary instruments or piezoelectric instruments (depending on the assignment to one of the two groups). Both surgical procedures involve complete closure of the wound by primary intention using sutures
  Arms: G1 - control group

SUMMARY:
To date, surgical therapy of MRONJ remains the therapy of choice while still in association with a medical approach. Surgical intervention aims to stop the progression of the pathology through the removal of the tissue macroscopically affected (resective surgery,sequestrectomy, debridement).

These surgical procedures are classically performed by the use of handpiece burs, but due to the advent of piezoelectric surgery in dentistry, a comparison of the two techniques is required

At present there are no randomized clinical trials designed to compare the postoperative discomfort of the two previously described techniques in the treatment of MRONJ. Therefore, the aim of this study is to evaluate the postoperative discomfort in a group of patients undergoing surgical therapy for MRONJ with piezoelectric instruments compared to a control group undergoing MRONJ surgical therapy with traditional rotary instruments.

METHODS This is a randomized clinical trial conducted in patients diagnosed with MRONJ who require surgical therapy.

Patients will be recruited and evaluated for a period of 24 months. Follow-up of patients enrolled in the study will last 12 months. Specifically, once patients diagnosed with MRONJ requiring surgical therapy are identified, surgery will be scheduled within 1 month, then follow-up visits will be conducted at 1, 2, 3 weeks and 3, 6, 12 months after surgery.

Patients enrolled and randomized into one of the two groups will all undergo necrotic bone removal surgery by the same operator with decades of experience in treating MRONJs. Marginal bone resection surgery will be performed using rotary or piezoelectric instruments. Both surgical procedures involve wound closure by first intention healing using sutures. Each bone block removed will undergo histologic examination for diagnostic confirmation of osteonecrosis. Postoperative instructions will be explained to patients, and sutures will be removed at 7 or 14 days after surgery.

Each patient will be asked for a 3D radiologic exam (CT or CBCT) at least 12 months after surgery in order to asses the

DETAILED DESCRIPTION:
Medicaiton-related osteonecrosis of the jaw (MRONJ) is defined as a drug-related adverse reaction characterized by progressive destruction and necrosis of the mandibular and/or maxillary bone in subjects exposed to treatment with drugs known to be at increased risk of disease, in the absence of previous radiation treatment. The first case of osteonecrosis was described in 2003 by Marx et al. in association with a specific group of drugs used in the treatment of skeletal system diseases: bisphosphonates, in particular the category of amino-bisphosphonates (i.e., zoledronate, pamidronate, alendronate) has been linked to the onset of MRONJ. However, from 2008, the first reports of MRONJ in association with other categories of drugs appeared: denosumab and targeted therapy as cancer treatment, such as bevacizumab, sunitinib, everolimus, etc. Bisphosphonates and denosumab are drugs used to treat osteometabolic (e.g. osteoporosis), oncological (e.g. bone metastases from solid tumors) and hematological diseases, available on the market in the form of oral or parenteral formulations (intravenous, intramuscular, subcutaneous). These drugs determine, through different mechanisms, an inhibition of osteoclastic activity and, consequently, an alteration of bone turnover. Target therapy are instead used only in the treatment of oncological diseases and mostly have an anti-angiogenic activity. The risk of onset of MRONJ varies mainly based on the type of drug administered, the administration route and the type of disease for which the intake was necessary; in particular, it has emerged that the risk is increased in case of intravenous administration and a higher cumulative dose, which is why cancer patients would seem to have a higher risk of developing MRONJ compared to subjects who use anti-resorbable drugs for osteo-metabolic diseases. The diagnostic process is complex and requires the integration of different clinical and radiological signs. In the past, the key element for the diagnosis of MRONJ was the presence of exposed necrotic bone inside the oral cavity, however in the literature it has emerged that a significant number of patients treated with these drugs present signs and symptoms, both in the initial and late phase, different from bone exposure alone. The diagnosis of MRONJ is structured according to the diagnostic work-up proposed by SICMF (Italian Society of Maxillo-Facial Surgery) - SIPMO (Italian Society of Oral Pathology and Medicine):

* Step 1: diagnostic suspicion deriving from the medical, dental and pharmacological history
* Step 2: differential diagnosis through identification of clinical signs (bad breath, odontogenic abscess, mandibular asymmetry, pain of dental and/or bone origin, exposure of necrotic bone, mucosal fistula, extra-oral fistula, hyperemia of the mucosa, failure to repair the alveolar mucosa after extraction, rapid onset of tooth mobility, preternatural mobility of the mandible, with or without preserved occlusion, paresthesia/dysesthesia of the lips, discharge from the nose, purulent discharge, spontaneous sequestration of bone fragments, trismus, swelling of the soft tissues), evaluation of pain and 1st level imaging (orthopantomography and/or intraoral radiography);
* Step 3: conclusive diagnosis through 2nd level imaging (CT Dentascan or Cone-Beam) These new diagnostic elements have allowed us to frame the pathology within a staging based on minor clinical signs and radiological signs. Reference is made to the staging proposed by SICMF - SIPMO. The importance of a correct diagnosis and therefore the inclusion of the pathology within a given stage lies in the variability and invasiveness of the therapeutic approach to MRONJ.

The treatment of MRONJ includes the possibility of medical and/or surgical therapy, although there is still no worldwide guidelines.

Medical therapy involves the use of drugs aimed at controlling the infection with the aim of stabilizing the clinical features by slowing the progression of the disease, but it is a very conservative approach that is unlikely to determine a complete resolution of the pathology. It consists of the association of an antiseptic therapy with chlorhexidine-based mouthwashes for disinfecting the oral cavity and an antibiotic therapy based on penicillins or in allergic patients quinolones, metronidazole, clindamycin and doxycycline.

Surgical therapy of MRONJ, however, remains the therapy of choice to date, although always in association with a medical approach. The surgical intervention, in fact, aims to stop the progression of the pathology through the removal of the tissue macroscopically involved in the disease until healthy bone tissue is reached.

The invasiveness of surgical techniques is strictly related to the staging and extension of MRONJ and, although there are no standard protocols, the aforementioned techniques can empirically be divided into:

* Resective surgery which involves the en bloc removal of the pathological bone until reaching the healthy vital tissue. It can be divided into segmental or marginal resective surgery if the intervention involves or does not involve the interruption of the anatomical continuity of the affected skeletal segment.
* Sequestrectomy which allows the surgical removal of a bone sequestration in the maxillary and/or mandibular area and is a simpler therapy than resective surgery, although there is difficulty in precisely identifying the microscopic limit between the bone involved in the disease and healthy tissue.
* Debridement which involves the surgical removal of necrotic bone tissue until a bleeding bone surface is identified. This procedure requires that the necrotic bone is not yet separated from the surrounding vital bone, otherwise it would be a sequestrectomy.

These surgical procedures are classically performed using burs mounted on a straight handpiece, but the advent of piezoelectric surgery in various areas of oral surgery has led us to the need for a comparison between the two techniques in the field of surgical treatment of MRONJ.

In the last 20 years, the use of ultrasonic vibrations has become routine for standard clinical applications in many fields of surgery, as it is able to reduce the risk of damage to the surrounding soft tissues and critical structures such as vessels and nerves during the osteotomy. Piezosurgery, in fact, would allow greater precision in cutting, protection of vascular-nervous structures and better visibility of the surgical field, compared to rotating instruments. These properties are determined by the fact that frequencies between 25-29 kHz are used, capable of determining a selective cut of mineralized tissues compared to soft tissues. According to some studies, moreover, piezoelectric bone surgery seems to be more efficient in the first phase of bone healing, inducing an early colonization of the residual bone by bone morphogenetic proteins, a greater control of inflammation and therefore a faster bone remodeling. Some authors have attributed the following limitations to this technique: prolonged operating time, learning difficulties and the risk of determining bone overheating in the case of excessive working pressure [9]. Consequently, there is no agreement, considering the available evidence, on which surgical technique represents the gold standard in the treatment of MRONJ, especially in reference to the perception of post-operative discomfort by the patient.

At present, to the best of the authors' knowledge, there are no randomized clinical studies aimed at comparing the post-operative discomfort of the two techniques previously described, in the treatment of MRONJ.

AIM The primary objective of this randomized controlled trial (RCT) is to evaluate postoperative pain and discomfort in a group of patients undergoing surgical therapy for MRONJ with piezoelectric instruments, using as a control a group of patients undergoing surgical therapy for MRONJ with traditional rotary instruments. Secondary objectives will focus on the evaluation of clinical healing of the site, operator discomfort, discomfort felt by the patient during the procedure, duration of the procedure and the occurrence of disease recurrence over the following 12 months. An additional objective of the study is the preoperative definition of a radiographic margin of bone resection associated with a lower rate of MRONJ recurrence by comparing the preoperative and postoperative three-dimensional radiographic examination (12 months after surgery).

Study design This is a prospective randomized and controlled parallel-group (1:1) superiority study. The study will be conducted blindly for the operator who collects the data and for the statistician, in order to ensure greater validity of the results. Randomization will occur after the flap lifting, preparatory to the surgical intervention of marginal resective surgery for the treatment of MRONJ. A randomization envelope will be opened at that moment, and the operator (the same for all the surgical procedures being studied) will proceed to complete the therapy with one or the other technique.

Study setting The study will be carried out at the UOC of General Dentistry and Orthodontics of the Fondazione Policlinico A. Gemelli - IRCSS. The care setting in which the patients enrolled in this study will be treated is of an outpatient type.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the information provided and to give free consent;
* Age greater than 18 years at the time of diagnosis;
* Diagnosis of stage 1 or stage 2 MRONJ, according to the SICMF-SIPMO classification [1];
* Need for surgical treatment of MRONJ.

Exclusion Criteria:

* Patients with a previous history of radiotherapy in the head and neck area;
* Patients with psychiatric disorders;
* Women of childbearing age
* Patients in stages of MRONJ other than stage 1 and 2;
* Patients undergoing retreatment of MRONJ;
* Patients with general medical contraindications for oral surgery procedures;
* Patients unable to attend the outpatient visits required by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
MRONJ healing | 12 months
  Evaluation of disease recurrence over the following 12 months: this evaluation will be performed clinically (absence of symptoms, absence of exposed bone in the oral cavity, and other minor clinical signs) and radiographically through a routinely required 3D radiographic exam (CBCT or CT).

SECONDARY OUTCOMES:
operators discomfort | at the end of surgery
  Assessment of operators discomfort during surgery by submitting a questionnaire at the end of surgery
ambient noise | during the surgery
  Assessment of the ambient noise level during the intervention with a Decibel detector (Protmex PT6708)
duration of the surgery | during the surgery
  Evaluation of the duration of the surgery (Chronometer) of the osteotomy
correlation between clinical parameters and patient's perception | 8 hours after surgery and then at 7 and 21 days after surgery
  Assess whether there is a correlation between clinical parameters of healing (modified Landry's Healing Index) and patient's subjective perception
Risk factors | 8 hours after surgery and then at 7 and 21 days after surgery
  Identify any risk factors associated with unfavorable postoperative course both in terms of clinical healing and subjective perception
postoperative discomfort OHIP | 8 hours after surgery and then at 7 and 21 days after surgery
  Assessment of postoperative discomfort of patients undergoing marginal resective surgery (OHIP-14). These questionnaires will be administered at 8 hours after surgery and then at 7 and 21 days after surgery.
postoperative discomfort - QoR | 8 hours after surgery and then at 7 and 21 days after surgery
  Assessment of postoperative discomfort of patients undergoing marginal resective surgery (QoR-15). These questionnaires will be administered at 8 hours after surgery and then at 7 and 21 days after surgery.
postoperative discomfort (NRS) | 8 hours after surgery and then at 7 and 21 days after surgery
  Assessment of postoperative pain (NRS-10). These questionnaires will be administered at 8 hours after surgery and then at 7 and 21 days after surgery.
Clinical Healing HI | after surgery at 7 and 21 days after surgery
  Assessment of clinical healing of sites undergoing marginal resective surgery using the modified Landry Healing Index

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lajolo, MD,DDS, Principal Investigator — Catholic University of Rome
Locations (1):
- Catholic University, Roma, Italy

REFERENCES:
- [Background] Marx RE. Pamidronate (Aredia) and zoledronate (Zometa) induced avascular necrosis of the jaws: a growing epidemic. J Oral Maxillofac Surg. 2003 Sep;61(9):1115-7. doi: 10.1016/s0278-2391(03)00720-1. No abstract available. PMID 12966493
- [Background] Mavrokokki T, Cheng A, Stein B, Goss A. Nature and frequency of bisphosphonate-associated osteonecrosis of the jaws in Australia. J Oral Maxillofac Surg. 2007 Mar;65(3):415-23. doi: 10.1016/j.joms.2006.10.061. PMID 17307586
- [Background] Yarom N, Fedele S, Lazarovici TS, Elad S. Is exposure of the jawbone mandatory for establishing the diagnosis of bisphosphonate-related osteonecrosis of the jaw? J Oral Maxillofac Surg. 2010 Mar;68(3):705. doi: 10.1016/j.joms.2009.07.086. No abstract available. PMID 20171493
- [Background] Ruggiero SL, Dodson TB, Fantasia J, Goodday R, Aghaloo T, Mehrotra B, O'Ryan F; American Association of Oral and Maxillofacial Surgeons. American Association of Oral and Maxillofacial Surgeons position paper on medication-related osteonecrosis of the jaw--2014 update. J Oral Maxillofac Surg. 2014 Oct;72(10):1938-56. doi: 10.1016/j.joms.2014.04.031. Epub 2014 May 5. PMID 25234529
- [Background] Colella G, Campisi G, Fusco V. American Association of Oral and Maxillofacial Surgeons position paper: Bisphosphonate-Related Osteonecrosis of the Jaws-2009 update: the need to refine the BRONJ definition. J Oral Maxillofac Surg. 2009 Dec;67(12):2698-9. doi: 10.1016/j.joms.2009.07.097. No abstract available. PMID 19925998
- [Background] El-Rabbany M, Sgro A, Lam DK, Shah PS, Azarpazhooh A. Effectiveness of treatments for medication-related osteonecrosis of the jaw: A systematic review and meta-analysis. J Am Dent Assoc. 2017 Aug;148(8):584-594.e2. doi: 10.1016/j.adaj.2017.04.002. Epub 2017 May 18. PMID 28527518
- [Background] Labanca M, Azzola F, Vinci R, Rodella LF. Piezoelectric surgery: twenty years of use. Br J Oral Maxillofac Surg. 2008 Jun;46(4):265-9. doi: 10.1016/j.bjoms.2007.12.007. Epub 2008 Mar 14. PMID 18342999